CLINICAL TRIAL: NCT01637064
Title: Acthar Dermatomyositis and Polymyositis Treatment
Brief Title: Dermatomyositis and Polymyositis Registry
Acronym: ADAPT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Phoenix Neurological Associates, LTD (Other)
Responsible Party: Sponsor
Other Study IDs: ADAPT
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Dermatomyositis; Polymyositis
Keywords: Myositis; Acthar treatment
MeSH Terms: conditions — Dermatomyositis; Polymyositis; Myositis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: None Retained — This is a retrospective and prospective study
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Acthar — Physicians will prescribe Acthar at their own discretion; however the recommended dose is 80 units subcutaneously twice a week.
  Other Names: ACTH

SUMMARY:
By creating a registry, physicians will have the opportunity to understand the clinical outcomes of Myositis patients treated with Acthar. Despite the availability of clinical exams, muscle biopsies, and other testing, it is surmised that there may be a more important classification of myositis that physicians are not diagnosing which could possibly lead to improper treatment due to inaccurate diagnosis. There may be several types of immune and inflammatory myositis (IIM) that do not fit well into the typical sub classifications of myositis.

DETAILED DESCRIPTION:
Retrospective and prospective data will be collected from physicians who have prescribed Acthar to myositis patients to determine what specific characteristics each patient has based on biopsy analysis, laboratory results, and clinical exams. Through biopsy analysis, subcategories of IIM will be determined and could illustrate which of these IIMs may be more responsive to Acthar therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85
2. Male or Female
3. Clinical or pathologic diagnosis of polymyositis or dermatomyositis
4. Capable of providing informed consent and complying with treatment regimen

Exclusion Criteria:

1. History of scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex
2. Recent surgery, history of or the presence of a peptic ulcer, congestive heart failure, uncontrolled hypertension, or sensitivity to proteins of porcine origin
3. Any other co-morbid condition which would make completion of the trial unlikely
4. If female, pregnant or breast-feeding; or, if of childbearing age, an unwillingness to use appropriate birth control

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All sites chosen are well-established universities, academic centers or private practices that specialize in neuromuscular diseases. These are physicians who have several myositis patients and who are prescribing or would prescribe Acthar to myositis patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Determining if Acthar treatment improves disease progression | 2 years
  To create and maintain a registry linking clinical information, dosing and clinical response in patients with refractory myositis and to determine if Acthar treatment improves disease progression

SECONDARY OUTCOMES:
Subgroups may predict response to Acthar therapy | 2 years
  To determine if there are different subgroups that can be defined myopathologically that may predict response to Acthar therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Todd D Levine, MD, Principal Investigator — Phoenix Neurological Associates, LTD; Petros Efthimiou, MD, Principal Investigator — New York Presbyterian Brooklyn Methodist Hospital; Ara Dikranian, MD, Principal Investigator — Ara Dikranian MD; Justine Malone, MD, Principal Investigator — Neurology INC; Rup Tandan, MD, Principal Investigator — University of Vermont
Locations (5):
- United States (5):
  - PNA Center for Neurological Research, Phoenix, Arizona
  - Ara Dikranian MD, San Diego, California
  - Neurology INC, Columbia, Missouri
  - New York Methodist Hospital, Brooklyn, New York
  - University of Vermont, Burlington, Vermont